CLINICAL TRIAL: NCT04561596
Title: Virtually Augmented Self Hypnosis: Randomized Controlled Trial in Peripheral Vascular Interventions
Brief Title: Virtually Augmented Self Hypnosis in Peripheral Vascular Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salah D. Qanadli, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Salah D. Qanadli, MD, PhD, Professor, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00728
Record Dates: First submitted 2020-09-09; First posted 2020-09-23 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Anxiety Postoperative; Pain, Postoperative; Vascular Access Site Pain
Keywords: Anxiety; Pain; Virtual reality; Virtual reality autohypnosis; Hypnosis; Non-pharmacological approaches
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Pain | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autohypnosis (Experimental): Use of virtual reality with head mounted display
  Interventions: Device: OnComfort autohypnosis
- Control (Other): Treatment as usual
  Interventions: Other: Treatment as usual, without the OnComfort autohypnosis system

INTERVENTIONS:
Device: OnComfort autohypnosis — Participant arrive in our day care clinic and is prepared as any other patient in interventional radiology. The investigator will collect the signed informed consent form and proceed to randomization.
  The participant will then fill the pre and post-operative anxiety and pain questionnaire.
  The percutaneous vascular procedure will be performed as usual except for the virtual reality mask and autohypnosis software that will run during the whole intervention.
  Pain and anxiolytic medication are provided if needed during the intervention. Immediately after the intervention, the participant will fill the post-operative anxiety and pain questionnaire. The participant will be instructed to report anxiety and pain felt during the intervention.
  A clinical visit at 3 month is conducted as part of the standard clinical protocol. The participant will fill a 3rd questionnaire about the remembered anxiety and pain during the intervention.
  Arms: Autohypnosis
Other: Treatment as usual, without the OnComfort autohypnosis system — The Participant arrive in our day care clinic and is prepared as any other patient in interventional radiology. The investigator will collect the signed informed consent form and proceed to randomization.
  The participant will then fill the pre and post-operative anxiety and pain questionnaire.
  The percutaneous vascular procedure will be performed as usual. Pain and anxiolytic medication are provided if needed during the intervention. Immediately after the intervention, the participant will fill the post-operative anxiety and pain questionnaire. The participant will be instructed to report anxiety and pain felt during the intervention.
  A clinical visit at 3 month is conducted as part of the standard clinical protocol. The participant will fill a 3rd questionnaire about the remembered anxiety and pain during the intervention.
  Arms: Control

SUMMARY:
The aim of our study is to compare patients anxiety and pain during percutaneous vascular interventions with and without virtual reality autohypnosis.

DETAILED DESCRIPTION:
The participants in the control group will be treated under local anesthesia, following the usual care protocols.

The participants in the experimental group will be treated under the same conditions, except that they will experience virtual reality autohypnosis during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* > 18 years
* Any indication for a percutaneous vascular interventional with a single vascular access (angiography, phlebography, arterial intervention, venous intervention) planned to be done under local anesthesia

Exclusion Criteria:

* No French language comprehension, deaf or visually impaired patient
* Inability to sign informed consent
* Need of sedative medication
* History of motion sickness
* History of psychiatric disease such as paranoia, schizophrenia, deep water phobia and dementia
* Patient does not tolerate the virtual reality mask during the pre operative visit at Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Per procedural anxiety. | Day 1 (Immediately after the peripheral vascular intervention)
  Per procedural anxiety, measured by the Spielberger Anxiety State Inventory in French (Gauthier and Bouchard, 1993).
  The Spielberger Anxiety State Inventory is a self questionnaire of 20 items, each item scores from 1 to 4. The result of the test is the sum of the 20 items, therefore the result ranges from 20 to 80. A high score is related to a high level of anxiety at the moment of the test.

SECONDARY OUTCOMES:
Per procedural pain. | Day 1 (Immediately after the peripheral vascular intervention)
  Per procedural pain, measured by the visual analog pain scale. The visual analog pain scale rates pain from 0 to 10, 0 being the least pain imaginable and 10 the maximal pain imaginable.
Remembered per procedural anxiety. | 3 months
  Remembered per procedural anxiety measured by the Spielberg Anxiety State Inventory in French (Gauthier and Bouchard, 1993).
  The Spielberger Anxiety State Inventory is a self questionnaire of 20 items, each item scores from 1 to 4. The result of the test is the sum of the 20 items, therefore the result ranges from 20 to 80. A high score is related to a high level of anxiety at the moment of the test.
Remembered per procedural pain. | 3 months
  Remembered per procedural pain will be measured by the visual analog pain scale.
  The visual analog pain scale rates pain from 0 to 10, 0 being the least pain imaginable and 10 the maximal pain imaginable.
Adverse events | Day 1
  Device deficiencies
Serious adverse events | Day 90
  Amputation, mesenteric or renal ischemia, and death

CONTACTS AND LOCATIONS:
Overall Officials: Salah Dine Qanadli, Prof. MD PhD, Study Director — Unil, CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gullo G, Rotzinger DC, Colin A, Frossard P, Gudmundsson L, Jouannic AM, Qanadli SD. Virtually Augmented Self-Hypnosis in Peripheral Vascular Intervention: A Randomized Controlled Trial. Cardiovasc Intervent Radiol. 2023 Jun;46(6):786-793. doi: 10.1007/s00270-023-03394-1. Epub 2023 Mar 21. PMID 36944851
- [Derived] Qanadli SD, Gudmundsson L, Gullo G, Ponti A, Saltiel S, Jouannic AM, Faouzi M, Rotzinger DC. Virtually Augmented Self-Hypnosis applied to endovascular interventions (VA-HYPO): Randomized Controlled Trial Protocol. PLoS One. 2022 Feb 23;17(2):e0263002. doi: 10.1371/journal.pone.0263002. eCollection 2022. PMID 35196310